CLINICAL TRIAL: NCT04026919
Title: OK en Casa - ZAINDOO an Online Support Program for Caregivers of People With Dementia, a Randomized Controlled Trial.
Brief Title: Online Support Program for Dementia Caregivers
Acronym: OKenCASA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Igone Etxeberria, Principal Investigator, University of the Basque Country (UPV/EHU)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00423
Record Dates: First submitted 2019-07-16; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Effect Increased

STUDY DESIGN:
Masking Description: The random assignment of the participants was carried out according to the following criteria: 1) Prepare an unpredictable sequence of random numbers; and, 2) Keep this sequence hidden until the assignment was carried out. To hide the sequence, the person in charge of the random assignment was maintained out of the recruitment and pre-treatment evaluation.
  The assignment was carried out controlling the following variables: sex, age (over or under 60 years), burden (score> 17 in the Reduced Zarit caregiver burden interview), attendance or not to the SENDIAN program (psychological support users) and / or support groups or non-users) of the primary caregiver and the level of dependence of the elderly person with dementia (mild / moderate or severe).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- to analyze the effectiveness of Ok en Casa Zaindoo (Experimental): The multicomponent online programme is composed of the components explained in the detailed study description:
  Interventions: Other: OK EN CASA-ZAINDOO

INTERVENTIONS:
Other: OK EN CASA-ZAINDOO — Intervention based on cognitive- behavioural techniques offered in an online format.

SUMMARY:
There are currently 50 million people in the world diagnosed with dementia. Due to the detrimental impact on the mental and physical health of family caregivers different online interventions have been developed in order to improve their well-being. In this paper, we describe the design of a randomized controlled trial aiming to study the impact of a multicomponent online program on primary and secondary caregivers of a person with dementia (PWD).

The experimental group will receive the intervention which is a multicomponent program based on different components, among others; online psychoeducation, training on psychological skills, a forum with other caregivers and interaction with a psychologist. Caregivers in the control group will follow their lifestyle.

More than 250 participants (primary and secondary caregivers) are expected to be recruited via several sources in the province of Guipuzcoa in Spain. The inclusion criteria for the primary caregiver are: a) being 18 years or older; b) being the primary caregiver of the PWD; c) more than 6 months caring; and d) give more than 1 hour of caregiving per day. The outcomes of this trial are caregiver burden (primary outcome), perceived health, depression and anxiety, social support, satisfaction with care and with the treatment and stress caused by the problem behaviour of the PWD (secondary outcomes).

DETAILED DESCRIPTION:
Aim: to analyze the effectiveness of a multicomponent online program on primary and secondary caregivers of a person with dementia.

Methods and analyses: The trial design is a two group randomized controlled trial to establish the effectiveness of an online support program. The experimental group will complete the program for 9 months and the control group will continue with their usual lifestyle. The objective is to examine the effect of this online support program on burden as primary outcome. Secondary outcomes of the study are social support, perceived health, anxiety, depression, satisfaction with caregiving, stress derived from the memory and behaviour problems of the person with dementia and satisfaction with treatment. The intervention will last for 9 months in total and includes two measurements, pre and post measure (9 months after) for the experimental and control group. The trial is set in Spain, concretely in The Basque Country.

OK en casa - Zaindoo: online support program for caregivers of persons with dementia. The multicomponent online programme is composed of the following components:

Assessment: In this section are placed the assessment tools that the caregiver must complet online before and after the intervention. The questionnaires collect information regarding the care context, health (perceived health, depression and anxiety), burden, satisfaction with care, family support and formal support (instrument created ad hoc).

My status: It offers information and feedback on the context of care, health and the socio-emotional status of the caregiver. It is composed of six blocks (context of care, health, burden, satisfaction with care, family support and formal support). The information offered to the caregiver is based on a system of colours that oscillates between green (optimal situation) and red (critical situation). Thus, and for each of the blocks indicated above, if the caregiver is in an optimal state or have few difficulties the green colour is shown. If has mild symptoms or difficulties in the care context the yellow colour is shown, the orange would represent moderate symptoms and difficulties and finally, the red colour is indicative of a critical socio-emotional situation or serious difficulties in the context of care. Likewise, a single colour is shown as a summary that reflects the general situation of the caregiver, respecting the order of the colours that have been explained above. The colour corresponding to each of the blocks and the one regarding the general situation is accompanied by a text that summarizes caregivers situation using a positive language.

PSYCHOSOCIAL INTERVENTION: Psychoeducational programme: In this section, the caregiver is recommended a personal plan of structured psychoeducational activities. These activities had been organized from lesser to greater difficulty and in their design and development the care phase in which the caregiver is has been taken into account (acquisition, consolidation or resolution). The activities are different depending on the type of caregiver: primary or secondary. The aim is to train the caregivers in psychological strategies and skills to face the care in the most optimal way possible (self-instructions, relaxation techniques, training in communication skills, problem behaviour management, emotion regulation). The activities are also aimed at focusing on the positive aspects related to care.

Online-training: In addition to the psychoeducational activities and based on an e-learning format, the caregiver is offered the possibility to make a personalized online training based on the evaluation made previously. These are videos with content created ad hoc for the study and dealing with various aspects related to the care of the person with dementia and the caregivers self-care.

Psychosocial support: It includes online psychosocial support with specialized psychologists. A total of 8 online support sessions are arranged, 6 of the appointments are set in advance and the caregiver is given the option of contacting another 2 times according to their own needs.

Social networking: each caregiver can interact with other caregivers through a chat. In addition, they can include reading material related to the care that can be discussed in the forum.

WALL: It is a space in which various messages are published daily, in some cases inspirational (i. e. motivating messages), in other cases reminder messages are sent to the caregiver (i. e. reminder of an appointment with the psychologist) and also auto -promotional (i. e. move the caregiver to do things for their own benefit). Messages of support sent by famous people or recognized by the community are also published, testimonies of other caregivers, and divulgation articles also appear. The main objective is to offer motivating social support and emotional support to the caregiver.

CARE TEAM AND CHAT: This is the place where the profile of each of the members of the care team is created, that is the primary and secondary caregivers of the person with dementia. In addition, a chat is included to exchange information about the cared person, for example, appointments with health personnel, social workers, incidents in care, medication modifications, patient's condition, etc.

ORGANIZATION: This element is set up to facilitate the care of the person with dementia. An appointment calendar is shown on the screen (doctors, nurse, social worker, lawyer, etc.). There is a repository where documents can be attached with the aim of facilitating communication between all the members of the care team. This is an organization system shared by the care team, so that both the primary caregiver and the secondary caregivers have access to the organization system.

POINTS PROGRAM: The caregiver receives a series of points for performing various actions, such as, for example, online training, etc. These points can be exchanged for various services related to health and self-care (for example, massages, tickets for a thalassotherapy center, discounts, etc.).

ACHIEVEMENT MARKER (1-15): Based on an intermittent reinforcement the caregiver reaches some achievements, but he does not always know what he has done to get it.

LEVEL MARKER: Indicates the level of the caregiver according to the progress he or she is making. It ranges between 1 (lower level) and 5 (higher level). In addition, informs about how much is missing to pass the level.

Randomization The random assignment of the participants was carried out according to the following criteria: 1) Prepare an unpredictable sequence of random numbers; and, 2) Keep this sequence hidden until the assignment was carried out. To hide the sequence, the person in charge of the random assignment was maintained out of the recruitment and pre-treatment evaluation.

The assignment was carried out controlling the following variables: sex, age (over or under 60 years), burden (score ≥ 17 in the Reduced Zarit caregiver burden interview), attendance or not to the SENDIAN program (psychological support users) and or support groups or non-users) of the primary caregiver and the level of dependence of the elderly person with dementia (mild- moderate or severe). Therefore, a stratified randomization was carried out, which is more appropriate than simple randomization when the sample size is not very large. The randomization unit were the families.

The precise randomization procedure consisted of ordering the participants according to the controlled variables and, by means of a sequence of random numbers, the participants were assigned to the treatment group or to the control group on the waiting list. Due to random it is possible that the size of the groups will be not exactly the same.

Procedure Sample recruitment Family caregivers of people with dementia were recruited via information letters and flyers through relevant institutions (San Sebastian City Council, basic social services, BetiOn (tele-assistance service of the Basque Government), social services of the Provincial Council of Gipuzkoa, health centers, pharmacies of Donostia, and the Association of Relatives and Friends of Persons with Alzheimer and other dementias of Guipuzcoa (AFAGI). Both the letters and the flyers provided a contact telephone associated with a call center in which calls were received from families interested in participating. The person in the call center answered the family's call, the possible questions they had, and if were interested to participate, the person in the call center collected the necessary data to check if they met with the inclusion and exclusion criteria. Afterwards the project team analyzed each case, and if complying with inclusion criteria the family was finally included in the study (primary caregiver and secondary caregivers).

Pre-Measurement It was performed online at the home of the caregivers with the support of students of the Social Work degree specifically trained to collect data. During this visit, informed consent was first collected and the pre-treatment evaluation was subsequently carried out using the evaluation protocol established. The students helped the caregivers to complete the evaluation protocol online (Tablet or Smartphone). It is hoped that they will learn to perform the evaluation without help on the next occasion.

ELIGIBILITY:
Inclusion Criteria:

* To be the main caregiver of the person with dementia
* To be over 18 years of age
* Provision of at least 6 months of care
* Provide at least one hour of care per day.

Exclusion Criteria:

* Having a contractual relationship for caring issues with the elderly person with dementia or with its family
* Have a disease that makes participation difficult during this pilot study (18 months)
* Not to have dementia.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Burden | Day 0, Month 0 and Day 0, Month 9
  Reduced Zarit burden scale (ZBI, Regueiro Pérez, Gómara & Ferreiro, 2007). It consists of 7 items that measures the perceived burden of caregivers via 5-point Likert scale items (0 = never, 1 = almost never, 2 = sometimes, 3 = many times, and 4 = almost always). This instrument establishes different degrees of overload depending on the score obtained. Scores lower than 17 are indicative that there is no overload, while scores higher than 17 indicate the existence of it.

SECONDARY OUTCOMES:
Memory and behavior problems | Day 0, Month 0 and Day 0, Month 9
  Memory and Behavior Problems Checklist (MBCL, Zarit & Zarit, 1982, translated by Izal & Montorio, 1994). This inventory consists of two subscales that measure the frequency of appearance of each problem and the stress caused to the caregiver. Each of these subscales consists of 30 items that are evaluated by a Likert-type scale with response options ranging from 0 to 4. In this study, the first 17 items that refer to problematic behaviors were applied.
Health status | Day 0, Month 0 and Day 0, Month 9
  collected by the following item: "In general, you would say that your health is very good, good, fair, bad or very bad". This item has been validated as a valid measure of the subjective perception of health in national and international studies.
  collected by the following item: "In general, you would say that your health is very good, good, fair, bad or very bad".
Anxiety and depression | Day 0, Month 0 and Day 0, Month 9
  The Hospital Anxiety and Depression Scale (Zigmond & Snaith, 1983). The tool includes 14 items and was designed for the evaluation of anxiety and depression in non-psychiatric outpatient hospital services. Seven items are related to anxiety and seven associated with depression, each scored between 0 (never) and 3 (almost all day). The authors recommended that a score above 8 on an individual scale should be regarded as a possible case and a score above 11 a probable case. It is a useful instrument validated in our environment (Quintana, Padierna, Esteban, Aróstegui, Bilbao, & Ruiz, 2003).
Social support | Day 0, Month 0 and Day 0, Month 9
  Family APGAR (Bellón, Delgado, Luna, & Lardielli, 1996). This scale shows the level of perceived dysfunctionality of a family unit assessed in a global way. The person evaluates each of the items using a Likert scale that oscillates between 0 (almost never) and 2 (almost always). The cut off points on the scale are the following: 0 to 2 points would indicate that there is a severe dysfunctionality among the family, between 3 and 6 would be slightly dysfunctional families, and finally, scores between 7 and 10 would indicate that it is a normo-functional family.
Satisfaction with care | Day 0, Month 0 and Day 0, Month 9
  The Caregiving Satisfaction Scale (CSS, Lawton, Kleban, Moss, Rovine & Glicksman, 1989, Spanish version of Lopez & Crespo, 2003). This scale measures the satisfaction of the caregiver from the caregiving situation. It consists of 6 items and the respondents are asked to rate each statement on a five-point scale ranging from 1 (strongly agree) to 5 (strongly disagree). Higher numbers reflect lesser satisfaction from the caregiving situation.
Satisfaction with the treatment | Day 0, Month 0 and Day 0, Month 9
  The Client Satisfaction Questionnaire (CSQ, Larsen, Attkinson, Hargreaves & Nguyen, 1979). This questionnaire will be administered to the caregivers in the experimental group at the end of the intervention program. Consists of a structured survey used to assess the level of satisfaction with the treatment. Items are scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction) with different descriptors for each response point. Total scores range from 8 to 32, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Igone Etxeberria, doctor, Principal Investigator — University of the Basque Country (UPV/EHU)
Locations (1):
- University of the Basque Country, San Sebastián, Guipuzcoa, Spain

IPD SHARING:
Plan to Share IPD: No